

## **OPERATe**

## **Consent Form**

If you are happy to participate please complete and sign the consent form below.

| | Activities | Initials |
|---|---|---|
| 1 | I confirm that I have read the attached information sheet (Version 2.0, Date 13/01/2025) for the above study and have had the opportunity to consider the information and ask questions and had these answered satisfactorily. | |
| 2 | I understand that my participation in the study is voluntary and that I am free to withdraw at any time without giving a reason and without detriment to myself. I understand that it will not be possible to remove my data from the project once it has been anonymised and forms part of the data set. | |
| 4 | I agree to take part on this basis. I understand that individuals from Manchester University NHS Foundation Trust will access my medical records to collect information for the study. I give permission for these individuals to have access to my records. | |
| 6 | I agree that any research publications can include direct quotes of my responses in anonymous format. | |
| 8 | I agree that any data collected may be included in anonymous form in publications/conferences presentations. | |
| 9 | I agree that any anonymised data collected may be made available to other researchers. | |
| 11 | I understand that data collected during the study may be looked at by individuals from The University of Manchester, Manchester University NHS Foundation Trust and/or regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my data. | |
| 12 | I understand that there may be instances where during the course of the research information is revealed which means the researchers will be obliged to break confidentiality and this has been explained in more detail in the information sheet. | |
| 13 | I agree to give the research team access to my personal wearable device token for collection of data. If you would like more general information on how researchers use data about patients, please visit: <a href="www.hra.nhs.uk/information-about-patients/">www.hra.nhs.uk/information-about-patients/</a> | |
| 14 | I agree to take part in this study. | |

The following activities are optional, you may participate in the research without agreeing to the following:

IRAS ID: 316796

Version 4.0 13/01/2025



| MAIN | 1824 reity of Manshorter |
|---|---|
| 15 | I agree that any pseudonymised, non-identifiable personal data collected may be made available to other researchers |
| 16 | I agree that the researchers may contact me in future about other research projects. |
| Optional Activities | |
| 3 | I agree to my GP being informed of my participation in this study. |
| Data Protection The personal information we collect and use to conduct this research will be processed in accordance with UK data protection law as explained in the Participant Information Sheet and the <a href="Privacy Notice for Research Participants">Privacy Notice for Research Participants</a> . | |
| By signing this consent form, I declare that I have provided accurate identity details (full name and electronic signature). | |
| Name of Participant Signature Date | |

1 copy of the consent form for the participant, 1 copy of the consent form for the research team (original) and, 1 copy of the consent form will be included in the patients notes.

Date

Signature

IRAS ID: 316796

Version 4.0 13/01/2025

Name of the person taking consent